CLINICAL TRIAL: NCT02420210
Title: Multicenter Phase II Study of the Bendamustine, Obinutuzumab, and Dexamethasone (BOD) Regimen in Un-fit Elderly ≥ 70 Years of Age Diffuse Large B-Cell Non-Hodgkin Lymphoma (DLBCL) Patients
Brief Title: Bendamustine, Obinutuzumab, and Dexamethasone in Older Patients With Diffuse Large B-cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trials was stopped early due to lack of funding.
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-1120; NCI-2015-00355 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB14-1120 (Other: University of Chicago Comprehensive Cancer Center); P30CA014599 (NIH)
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Results first posted 2018-03-14 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Bendamustine Hydrochloride; obinutuzumab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (bendamustine, obinutuzumab, dexamethasone) (Experimental): Patients receive bendamustine hydrochloride IV over 30 minutes on days 1 and 2, obinutuzumab IV over 4 hours on days 1 or 2, 8, and 15 (on both days 1 and 2 in course 1 only), dexamethasone PO daily on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bendamustine Hydrochloride; Biological: Obinutuzumab; Drug: Dexamethasone; Other: Quality-of-Life Assessment; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Bendamustine Hydrochloride — Given IV
  Other Names: Ribomustin; SyB L-0501; Treanda
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA101; Gazyva; R7159; RO 5072759
Drug: Dexamethasone — Given PO
  Other Names: DM
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well bendamustine hydrochloride, obinutuzumab, and dexamethasone work in treating older patients with diffuse large B-cell lymphoma. Drugs used in chemotherapy, such as bendamustine hydrochloride and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as obinutuzumab, may find cancer cells and help kill them. Giving bendamustine hydrochloride, obinutuzumab, and dexamethasone may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the overall response rate (ORR; complete responders [CR] + partial responders [PR]) using the Cheson et al parameters of this novel combination regimen.

SECONDARY OBJECTIVES:

I. Assess the feasibility of incorporating prospective geriatric assessments in patients >= 70 years of age diagnosed with diffuse large B-cell lymphoma (DLBCL) and treated in a multi-center setting.

II. Quality of life (QOL) based on Functional Assessment of Cancer Therapy-Lung (FACT-L) scale on all enrolled patients.

III. Progression-free survival (PFS) at 2 and 3 years. IV. Overall survival (OS) at 2 and 3 years.

OUTLINE:

Patients receive bendamustine hydrochloride intravenously (IV) over 30 minutes on days 1 and 2, obinutuzumab IV over 4 hours on days 1 or 2, 8, and 15 (on both days 1 and 2 in course 1 only), dexamethasone orally (PO) daily on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 40 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed DLBCL, cluster of differentiation (CD)20 positive by flow or immunohistochemistry (IHC); transformed DLBCL is allowed as long as no prior therapy has been given
* No prior therapy for DLBCL, except =< 1 week of corticosteroids given on an emergent basis or as a temporizing measure (pre-phase where indicated by the treating physician)
* Measurable disease by computed tomography (CT), magnetic resonance imaging (MRI), and/or positron emission tomography (PET) with at least one target lesion measuring 1.5 cm or larger
* Patients must be considered ineligible for rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate and prednisone (R-CHOP) standard therapy; to be ineligible for R-CHOP, patients must meet at least one of the following criteria are met:

  * Prior anthracycline therapy for other malignancies or other disorders whereby if additional anthracyclines are given for DLBCL, the maximum lifetime allowable dose will be exceeded
  * Meeting the geriatric criteria of ineligibility for standard R-CHOP if one of the following criteria is present:

    * Three or more organ systems with a score of 3 or any 1 organ system with a score of 4 (using the Cumulative Illness Rating Scale for Geriatrics, [CIRS-G])
    * Score of 3 or above on the Vulnerable Elders Survey (VES-13)
    * Score of =< 9 in the short physical performance battery (SPPB)
    * Presence of a significant geriatric syndrome (dementia, delirium, falls, incontinence, malnutrition, and severe osteoporosis) in the past year prior to diagnosis
    * Any abnormality in performing activities of daily living (ADLs) or instrumental activities of daily living (IADLs)
* Absolute neutrophil count (ANC) >= 1.5 unless cytopenias are related to bone marrow involvement with disease
* Hemoglobin >= 7 g/dl unless cytopenias are related to bone marrow involvement with disease
* Platelets >= 75,000 unless cytopenias are related to bone marrow involvement with disease
* Glomerular filtration rate (GFR) > 30 using Cockcroft-Gault formula
* Total bilirubin =< 3 times the upper limit of normal unless hepatic dysfunction is related to liver involvement with disease
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 5.0 times the upper limit of normal unless hepatic dysfunction is related to liver involvement with disease
* Alkaline phosphatase =< 5.0 times the upper limit of normal unless hepatic dysfunction is related to liver involvement with disease
* The ability to understand and sign a written informed consent

Exclusion Criteria:

* Prior therapy for DLBCL
* Other non-Hodgkin lymphoma (NHL) histologies
* Known central nervous system (CNS) involvement
* Known human immunodeficiency virus (HIV) or human T-lymphotropic virus, type I (HTLV-I) positive status
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver involvement with NHL or stable chronic liver disease per treating investigator assessment)
* Treatment with any known non-marketed drug substance or experimental therapy within 4 weeks prior to enrollment, or currently participating in any other interventional clinical study for NHL or any other illness (except observational and registry trials)
* Other past or current malignancy; subjects who have been free of malignancy for at least 3 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma (any site) are eligible; women with a history of cervical cancers are allowed
* Chronic or current infectious disease requiring systemic antibiotics, antifungal (excluding antifungals given for nail-beds infections), or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active hepatitis C
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae
* Positive hepatitis serology:

  * Hepatitis B virus (HBV): patients with positive serology for hepatitis B defined as positivity for hepatitis B surface antigen (HBsAg) or anti-hepatitis B core antibody (HBc); patients who are positive for anti-HBc may be considered for inclusion in the study on a case-by-case basis if they are hepatitis B viral deoxyribonucleic acid (DNA) negative and are willing to undergo ongoing HBV DNA testing by real-time polymerase chain reaction (PCR); patients with positive serology may be referred to a hepatologist or gastroenterologist for appropriate monitoring and management
  * Hepatitis C (hepatitis C virus [HCV]): patients with positive hepatitis C serology unless HCV ribonucleic acid (RNA) is confirmed negative and may be considered for inclusion in the study on a case-by-case basis
* Positive serology for hepatitis C (HC) defined as a positive test for hepatitis C antibody (HCAb)
* Inability to comply with study or follow-up testing and procedures
* Prior radiotherapy is allowed if it was given for low-grade lymphoma before transformation in those with transformed NHL and as long as no chemotherapy was administered in conjunction with radiation
* Any patient receiving a live vaccine must allow a 4-week interval before starting treatment on this study
* Known hypersensitivity to mannitol
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy or a known hypersensitivity to any of the other study drugs
* Major surgery within 4 weeks from cycle # 1
* Fertile men or women of childbearing potential unless 1) surgically sterile or 2) using an adequate measure of contraception such as oral contraceptives, intrauterine device, or barrier method of contraception in conjunction with spermicidal jelly
* Effective contraception is required while receiving obinutuzumab; for women, effective contraception is required to continue for >= 12 months after the last dose of obinutuzumab; for men, effective contraception is required to continue for 3 months after the last dose of obinutuzumab treatment
* Vaccination with a live vaccine a minimum of 28 days prior to the start of treatment

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Cohen, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Bendamustine, Obinutuzumab, Dexamethasone)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Bendamustine, Obinutuzumab, Dexamethasone)
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 89.5 [88 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: ORR (PR + CR) Using the Cheson et al Parameters
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bendamustine, Obinutuzumab, Dexamethasone)
Number analyzed (Participants) | 2
Participants | 2

2. Secondary Outcome: Feasibility, Defined as Completing All Required Geriatric Assessments Where Applicable Per the Protocol in 80% or More of the Enrolled Eligible Patients
Time Frame: Up to 40 months
Population: Funding for study was withdrawn after two patients were enrolled. Secondary outcomes not collected.
Arm/Group | Treatment (Bendamustine, Obinutuzumab, Dexamethasone)
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Survival analyses will be performed according to Kaplan and Meier methods. Prognostic factors that predict favorable outcomes and responses will be evaluated in both univariate and multivariate analyses using Cox proportional hazards regression for possible indicator of better OS. OS will also be stratified for bulky versus non-bulky disease comparisons (defined as any site with more than 5 cm in largest diameter).
Time Frame: From date of study entry (date of first treatment) until death from any cause, assessed at 2 years
Population: Funding for study was withdrawn after two patients were enrolled. Secondary outcomes not collected.
Arm/Group | Treatment (Bendamustine, Obinutuzumab, Dexamethasone)
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival (OS)
Description: as for outcome 3
Time Frame: From date of study entry (date of first treatment) until death from any cause, assessed at 3 years
Population: Funding for study was withdrawn after two patients were enrolled. Secondary outcomes not collected.
Arm/Group | Treatment (Bendamustine, Obinutuzumab, Dexamethasone)
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression Free Survival
Description: Kaplan-Meier analysis will be performed. Prognostic factors that predict favorable outcomes and responses will be evaluated in both univariate and multivariate analyses using Cox proportional hazards regression for possible indicator of better PFS.
Time Frame: From date of study entry (date of first treatment) until progression, secondary malignancy, or death from any cause, assessed at 2 years
Population: Funding for study was withdrawn after two patients were enrolled. Secondary outcomes not collected.
Arm/Group | Treatment (Bendamustine, Obinutuzumab, Dexamethasone)
Number analyzed (Participants) | 0

6. Secondary Outcome: Incidence of Toxicity Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Adverse events will be tabulated by type and grade.
Time Frame: Up to 30 days following the last administration of study treatment
Population: Funding for study was withdrawn after two patients were enrolled. Secondary outcomes not collected.
Arm/Group | Treatment (Bendamustine, Obinutuzumab, Dexamethasone)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Quality of Life Assessed Using the Functional Assessment of Cancer Therapy (FACT)-L Scale
Time Frame: Up to 18 weeks (at end of study treatment)
Population: Funding for study was withdrawn after two patients were enrolled. Secondary outcomes not collected.
Arm/Group | Treatment (Bendamustine, Obinutuzumab, Dexamethasone)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Treatment (Bendamustine, Obinutuzumab, Dexamethasone)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Bendamustine, Obinutuzumab, Dexamethasone) (N=2)
Anorexia (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Bendamustine, Obinutuzumab, Dexamethasone) (N=2)
White blood cell decreased (Investigations) | 1
Upper resipiratory infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes